CLINICAL TRIAL: NCT03082989
Title: Prospective Study Evaluating the Routine Standard Use of Fractional Flow Reserve and Disagreement With Guideline Recommendations: a Nationwide Study
Brief Title: Evolving Routine Standards in Intracoronary Physiology
Acronym: ERIS
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Società Italiana di Cardiologia Invasiva (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Associate Professor, University Hospital of Ferrara
Other Study IDs: 110109
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fractional flow reserve performed: consecutive patients with ischemic heart disease and clinical indication to coronary artery angiography where the operator decided to use fractional flow reserve to drive the revascularization
  Interventions: Device: fractional flow reserve performed
- fractional flow reserve not performed: consecutive patients with ischemic heart disease and clinical indication to coronary artery angiography and satisfying prespecified criteria where the operator decided to not use fractional flow reserve to drive the revascularization
  Interventions: Other: fractional flow reserve not performed

INTERVENTIONS:
Device: fractional flow reserve performed — assessing fractional flow reserve to drive revascularization
  Groups: fractional flow reserve performed
Other: fractional flow reserve not performed — description of the main reasons leading the operator to not use fractional flow reserve to drive the coronary revascularization
  Groups: fractional flow reserve not performed

SUMMARY:
Italy is the European country with the minor penetration of FFR as compared to the number of percutaneous coronary intervention.

Accordingly, the Società Italiana di Cardiologia Invasiva (SICI-GISE) conceived and promoted a prospective nationwide study to describe the patterns of the use of FFR in an unselected real-world population and to to assess the reasons, on clinical decision making, driving operators in the use or not of the FFR.

DETAILED DESCRIPTION:
Fractional flow reserve (FFR) has been validated as a reliable surrogate for inducible ischemia, supporting its use during invasive procedures for functional assessment of coronary lesions. Landmark randomized trials have demonstrated that deferral of nonsignificant lesions based on FFR is not only safe, but also that FFR-guided revascularization is associated with a better clinical outcome up to 2 years, when compared with standard angiography.

In spite of the overwhelming evidence of its potential clinical and economic benefits and strong guideline recommendation, the adoption of FFR in the real-world is perceived to vary significantly. Reasons for this disparity are several, but most operators still do rely the most on angiographic eye-balling to decide on the functional significance of coronary lesions and the need for revascularization.

Italy is the European country with the minor penetration of FFR as compared to the number of percutaneous coronary intervention.

Accordingly, the Società Italiana di Cardiologia Invasiva (SICI-GISE) conceived and promoted a prospective nationwide study to describe the patterns of the use of FFR in an unselected real-world population and to to assess the reasons, on clinical decision making, driving operators in the use or not of the FFR.

ELIGIBILITY:
Inclusion Criteria:

FRACTIONAL FLOW RESERVE PERFORMED GROUP

* age >18 years
* written consent
* assessment with FFR of at least one coronary lesion

FRACTIONAL FLOW RESERVE NOT PERFORMED GROUP

* age >18 years
* written consent
* absence of assessment with FFR of at least one coronary lesion

  + at least one of the following criteria
  1. stable coronary artery disease, absence of non-invasive stress test, evidence of coronary lesions between 50%-90% (visual estimation or quantitative coronary analysis)
  2. stable coronary artery disease, presence of non-invasive stress test, evidence of coronary lesions between 50%-70% (visual estimation or quantitative coronary analysis)
  3. acute coronary syndrome, culprit lesion not identifiable or coronary lesions different from the culprit between 50%-70% (visual estimation or quantitative coronary analysis)

     Exclusion Criteria:
* written consent denied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients with ischemic heart disease and clinical indication to coronary artery angiography
Sampling Method: Non-Probability Sample
Enrollment: 1858 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
agreement with current guidelines | intra-procedure
  percentage of patients receiving a FFR assessment in agreement with current guidelines

SECONDARY OUTCOMES:
reasons leading to FFR disuse | intra-procedure
  description of the main reasons leading operator to prefer not assessment of coronary

CONTACTS AND LOCATIONS:
Overall Officials: Marco Luciano Rossi, MD, Principal Investigator — Humanitas, Rozzano (MI); Giulio Stefanino, MD, Principal Investigator — Humanitas, Rozzano (MI); Matteo Tebaldi, MD, Principal Investigator — AOU Ferrara; Gianluca Campo, MD, Principal Investigator — AOU Ferrara; Massimo Fineschi, MD, Principal Investigator — AOU Siena; Giuseppe Musumeci, MD, Principal Investigator — AOU Cuneo
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tebaldi M, Biscaglia S, Fineschi M, Musumeci G, Marchese A, Leone AM, Rossi ML, Stefanini G, Maione A, Menozzi A, Tarantino F, Lodolini V, Gallo F, Barbato E, Tarantini G, Campo G. Evolving Routine Standards in Invasive Hemodynamic Assessment of Coronary Stenosis: The Nationwide Italian SICI-GISE Cross-Sectional ERIS Study. JACC Cardiovasc Interv. 2018 Aug 13;11(15):1482-1491. doi: 10.1016/j.jcin.2018.04.037. Epub 2018 May 23. PMID 29803695